CLINICAL TRIAL: NCT00397189
Title: A Double-blind, Parallel Group, Randomised, Placebo Controlled Study of Efficacy and Safety of Circadin® 2 mg in the Treatment of Insomnia Patients With Low Endogenous Melatonin
Brief Title: Efficacy and Safety of Circadin® 2 mg in the Treatment of Primary Insomnia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurim Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU 112006
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Results first posted 2011-03-28 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Primary Insomnia
Keywords: Primary insomnia as defined by DSM IV criteria
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Circadin (Experimental)
  Interventions: Drug: Circadin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo circadin

INTERVENTIONS:
Drug: Circadin — Prolonged release melatonin 2 mg
  Other Names: ATC code: N05CH01
  Arms: Circadin
Drug: placebo circadin — placebo circadin tablets
  Arms: placebo

SUMMARY:
This is a randomised, placebo controlled study to evaluate the efficacy of a 3 week treatment period with Circadin® 2 mg in shortening sleep latency in patients with primary insomnia aged 18-80 with melatonin deficiency.

DETAILED DESCRIPTION:
Studies throughout the world have shown that insomnia is a common complaint that occurs in 10-50% of the population depending on age, sex and country. Among the wide variety of available treatments of sleep disturbances, the most commonly prescribed hypnotics are the benzodiazepines (BZD) and non-BZD hypnotics.

However, these hypnotics were often associated with rebound, dependency, tolerance, higher risk of falls mainly in the elderly population, anterograde memory disturbances and increased risk for motor accidents the next day.

In response to the unmet clinical need for a safe and efficacious alternative treatment for primary insomnia, that in addition to treating quantitative sleep problems, would improve sleep quality and daytime functioning, a clinical development program on melatonin for the treatment of primary insomnia was initiated.

This study is conducted using a randomised, double-blind, placebo controlled parallel group design, after a single-blind placebo period. Primary insomnia patients aged 18-80 will be screened for entry into the study.

After the initial 3 weeks double-blind treatment period, patients will be given the option to enter a six-month double-blind continuation study.

Primary parameter is sleep latency, secondary parameter is sleep maintenance. Exploratory parameters are total sleep time, sleep quality, morning alertness and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and aged 18-80 years.
* Are willing to take a 6-SMT level evaluation test.
* Suffering from primary insomnia according to DSM-IV. criteria (307.42 primary insomnia, Appendix 24.3) .
* Sleep latency of at least 20 minutes.
* Have not been using benzodiazepines (BZD) and non-BZD hypnotics for the past 2 weeks or more.
* Have not been using psychotropic treatments for the past 3 months or more.
* Are stabilized on non-psychotropic treatments for more than 1 month.
* Are willing to sign a written informed consent to participate in the study.

Exclusion Criteria:

* Use of benzodiazepines or other hypnotics (including psychotropic treatments) during the study and preceding two weeks.
* Alcohol intake more than 30 g of pure alcohol per day and any intake after lunch-time.
* Pharmacological immunosuppression.
* Participation in a clinical trial with any investigational agent within two months prior to study enrollment.
* According to DSM IV, subjects belonging to the following groups are excluded: 780.59 (breathing related sleep disorder); 307.45 (circadian rhythm sleep disorder); 307.47 (dyssomnia not otherwise specified); 780.xx (sleep disorder due to general medical condition).
* Severe neurological, psychiatric disorders (especially psychosis, anxiety and depression) and alcoholism.
* Other serious diseases that could interfere with patient assessment.
* Pregnant or breast feeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 930 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon M Crawford, MBChB, Principal Investigator — CPS Research
Locations (1):
- CPS Research, Glasgow, United Kingdom

REFERENCES:
- [Derived] Wade AG, Crawford G, Ford I, McConnachie A, Nir T, Laudon M, Zisapel N. Prolonged release melatonin in the treatment of primary insomnia: evaluation of the age cut-off for short- and long-term response. Curr Med Res Opin. 2011 Jan;27(1):87-98. doi: 10.1185/03007995.2010.537317. Epub 2010 Nov 24. PMID 21091391
- [Derived] Wade AG, Ford I, Crawford G, McConnachie A, Nir T, Laudon M, Zisapel N. Nightly treatment of primary insomnia with prolonged release melatonin for 6 months: a randomized placebo controlled trial on age and endogenous melatonin as predictors of efficacy and safety. BMC Med. 2010 Aug 16;8:51. doi: 10.1186/1741-7015-8-51. PMID 20712869

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient entered the study on 24 October 2006 and the last patient completed the study (safety follow up) on 2 December 2008 (last patient completed the last visit on 24 October 2008).
Pre-assignment Details: 930 patients were enrolled into the study and entered the run-in period; 139 of these patients were discontinued during the run-in period. The main reasons for discontinuation from the run-in were unwillingness to continue and ineligible to continue. Treatment periods were 3 weeks double-blind (DB) (1:1) and extension period 26 weeks DB (3:1)
Groups:
- Circadin: Prolonged release melatonin 2 mg. Tablets should be taken 1-2 hours before going to bed.
- Placebo: Identical tablets to Circadin. Tablets should be taken 1-2 hours before going to bed.
Period: 3 Weeks Period
Arm/Group | Circadin | Placebo
Started | 394 | 395
Completed | 373 (out of 373, 360 were included in the ITT population detailed in the Baseline Characteristics.) | 373 (out of 373, 362 were included in the ITT population detailed in the Baseline Characteristics)
Not Completed | 21 | 22
Not completed — Lost to Follow-up | 5 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 13 | 9
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 0 | 3
Not completed — Other | 0 | 2
Period: Extension Period
Arm/Group | Circadin | Placebo
Started | 534 (Not all completers continued to extension as only patients who wished to proceed were randomized.) | 177 (Please note randomization ratio in extension is 3:1)
Completed | 421 | 134
Not Completed | 113 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Circadin | Placebo | Total
Number analyzed (Participants) | 360 | 362 | 722
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 223 | 218 | 441
  >=65 years | 137 | 144 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10) | 61.5 (10.5) | 61.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 253 | 244 | 497
  Male | 107 | 118 | 225
Region of Enrollment [Number; unit: participants]
  United Kingdom | 360 | 362 | 722

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in Subjective Sleep Latency.
Description: Sleep latency (SL) after 3 weeks of treatment was assessed by Patient Daily Sleep Diary (National sleep foundation sleep diary). The patients reported subjectively of their SL. The Sleep Diary question 3 (SL) was summarised at baseline (end of the two-week run-in period) and after three weeks double-blind treatment (actual and change from baseline) for each treatment group using descriptive statistics. At each visit, the mean of the seven days prior to the visit were used. For each treatment group, the mean score at visit 3 was compared, adjusting for the visit 2 score. An ANCOVA model was used. Lower score indicates reduction in sleep latency and thus considered improvement
Time Frame: Baseline and 3 weeks
Population: Pre-planned analysis on ITT population age 65-80
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Circadin | Placebo
Number analyzed (Participants) | 137 | 144
minutes | -19.1 (47.3) | -1.7 (47.8)
Statistical Analysis 1: Comparison: Circadin vs Placebo; The analysis was a comparison of sleep latency as measured by the sleep diary at Visit 3 in the ITT 65-80 population, using a linear regression model with terms for treatment (Circadin® 2mg vs. Placebo) and baseline sleep latency; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = -15.6, 95% CI 2-sided [-25.3 to -6], Standard Deviation 47

2. Secondary Outcome: The Change From Baseline in Subjective Sleep Maintenance.
Description: Sleep maintenance as measured by number of awakening (NOA) after 3 weeks of treatment was assessed by Patient Daily Sleep Diary (National sleep foundation sleep diary). The patients reported subjectively of their NOA. The Sleep Diary question 4 (NOA) was summarized at baseline (end of the two-week run-in period) and after three weeks double-blind treatment (actual and change from baseline) for each treatment group using descriptive statistics. At each visit, the mean of the seven days prior to the visit were used. For each treatment group, the mean score at visit 3 was compared, adjusting for the visit 2 score. An ANCOVA model was used. Lower score indicates less awakenings and thus considered improvement.
Time Frame: 3 weeks
Measure: Mean (95% Confidence Interval); unit: Awakenings
Arm/Group | Circadin | Placebo
Number analyzed (Participants) | 137 | 144
Awakenings | -0.24 [-0.33 to 0] | -0.09 [-0.33 to 0]

ADVERSE EVENTS:
Time Frame: 37 weeks (2 weeks baseline, 3 weeks double-blind, 26 weeks double-blind extension period and 2 weeks run-out,AEs were to be reported for up to 30 days after stopping study medication )
Description: The safety variables were assessed at each visit and included spontaneously reported adverse events (AEs); unusual events and AEs recorded by the investigator
Arm/Group | Circadin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/394 | 3/395
Other Adverse Events (participants affected / at risk) | 32/394 | 42/395
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Circadin (N=394) | Placebo (N=395)
cellulitis (Infections and infestations) | 1 (1) | 0 (0)
chest pain (General disorders) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Circadin (N=394) | Placebo (N=395)
nasopharyngitis (Infections and infestations) | 13 | 16
upper respiratory tract infection (Infections and infestations) | 8 | 8
headache (Nervous system disorders) | 11 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less